CLINICAL TRIAL: NCT02129738
Title: Is Reuse of Intermittent Urethral Catheters Safe and Preferred? A Prospective, Observational Study Evaluating Reuse of Catheters and Switch to Single-use.
Brief Title: Reuse of Intermittent Urethral Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LOF-0028
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Intermittent Urethral Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LoFric (Experimental): LoFric catheters
  Interventions: Device: LoFric catheters

INTERVENTIONS:
Device: LoFric catheters — LoFric single use catheters to be used 4-6 times daily for 4 weeks.

SUMMARY:
The purpose of this study is to investigate and document real life safety and satisfaction of re-use of urethral catheters for intermittent self catheterization. The study will collect re-used catheters from included patients and compare those to a control group with regard to bacterial contamination and mechanical properties. A four week prospective evaluation will follow where the patients will be given catheters intended for single-use.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Female and/or male aged 18 years and over
* Intermittent self-catheterization as primary bladder management method, defined as a normal catheterization frequency of at least 4 times daily
* Reuse of the same silicon, rubber (latex) or plastic (e.g. vinyl, PVC) catheter
* Accustomed intermittent catheterization user, defined as intermittent catheterization use for at least 3 months
* Able to use catheters of size:

  40 cm, CH12 or CH14; 16'', FR12 or FR14; 15 cm, CH10 or CH12; 6'', FR10 or FR12;

Exclusion Criteria:

* Antibiotic treatment within 4 weeks prior study inclusion
* Drug or alcohol abuse or other disease of addiction
* Immunocompromising diseases or medications
* Known urological/renal anatomical abnormalities with potential impact on subject´s compliance as judged by the investigator
* Diagnosis of severe fecal incontinence that may compromise study participation as judged by the investigator
* Involvement in the planning and conduct of the study (applies to both Wellspect HealthCare staff and staff at the study site)
* Previous enrollment in the present study
* Simultaneous participation in another clinical study that may interfere with the present study, as judged by the investigator
* Severe non-compliance to protocol as judged by the investigator and/or Wellspect HealthCare

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-06-20 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Proportion of catheters with bacterial contamination (Y/N) | At Baseline (Visit 1)
  Proportion of catheters with bacterial contamination verified by culturing/incubation and visual inspection by Scanning Electron Microscope (SEM).

SECONDARY OUTCOMES:
Bacterial quantification by incubation. | At Baseline (Visit 1)
Pathogen identification by incubation. | At Baseline (Visit 1)
Material properties and bacteria/particle/tissue visualization by SEM. | At Baseline (Visit 1)
Presence of reuse found in medical records, patient reported questionnaires and patient interviews. | At Baseline (Visit 1) and at 4 weeks (Visit 2)
Bacterial level in urine sample | At Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bonne Lee, Dr, Principal Investigator — Prince of Wales Hospital, Randwick, Australia; Diane Newman, Professor, Principal Investigator — University of Pennsylvania, Philadelphia, US
Locations (7):
- United States (3):
  - North Idaho Urology, Coeur d'Alene, Idaho
  - University of Pennsylvania, Penn Urology, Philadelphia, Pennsylvania
  - Froedtert Medical College and Specialty Clinic, Milwaukee, Wisconsin
- Australia (4):
  - Royal Rehab, Ryde, New South Wales
  - Prince of Wales Hospital Spinal Unit, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Caulfield Hospital, Spinal Rehabilitation Unit, Melbourne, Victoria

REFERENCES:
- [Derived] Newman DK, New PW, Heriseanu R, Petronis S, Hakansson J, Hakansson MA, Lee BB. Intermittent catheterization with single- or multiple-reuse catheters: clinical study on safety and impact on quality of life. Int Urol Nephrol. 2020 Aug;52(8):1443-1451. doi: 10.1007/s11255-020-02435-9. Epub 2020 Mar 14. PMID 32172456